CLINICAL TRIAL: NCT01935518
Title: A Historical Placebo Controlled Screening Trial of Safety and Efficacy of Fasudil in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: A Clinical Trial of Safety and Efficacy of Fasudil in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Fan Dongsheng, Chairman of the department of neurology of Peking University Third Hospital, Peking University Third Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUTH-2013121
Record Dates: First submitted 2013-09-01; First posted 2013-09-05 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — fasudil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fasudil (Experimental): All the patients will take the fasudil treatment for 14 days (30mg twice a day, intravenous). 3 months later they will repeat the treatment mentioned before.
  Interventions: Drug: Fasudil

INTERVENTIONS:
Drug: Fasudil — All the patients will take the fasudil treatment for 14 days (30mg twice a day, intravenous). 3 months later they will repeat the treatment mentioned before.

SUMMARY:
This study will examine whether fasudil is effective and safe in treating patients with amyotrophic lateral sclerosis (ALS).

DETAILED DESCRIPTION:
This is an open labeled, single center clinical study with placebo of historical researches as control. 10 patients will be enrolled in the study. The basic treatment is riluzole, 50mg twice a day. For the procedure, patients will take fasudil treatment for 14 days (30mg twice a day, intravenous). 3 months later, patients will repeat the fasudil treatment. All the patients will be followed up for 6 months. The primary outcome was the decline rate of ALSFRS-R. The secondary outcomes are the survival time, endpoint time(death, tracheotomy and continuous ventilator-dependent), forced vital capacity (FVC), the short form health survey (SF-36), evaluation of cognitive function (verbal fluency and Frontal Behavioral Inventory Scale) and safety.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of laboratory-supported probable, probable, or definite ALS
* Age: 18-70 years
* Disease duration: 3-36 months
* Forced vital capacity: at least 60% of predicted
* ALSFRS-R: at least 30, respiratory items: at least 10
* Decline of ALSFRS-R in the last 3 months before enrollment: 1-8
* Must take riluzole, on a stable dose for at least 30 days prior to baseline visit with no serious side effects. They must continue the riluzole treatment for at least 6 months after enrollment.
* Patients of childbearing potential must be using an effective method of birth control
* Willing and able to give informed consent

Exclusion Criteria:

* Familial ALS
* Pregnant or nursing women
* Patients after tracheotomy or continuous ventilator-dependent (time with non-invasive ventilator more than 22 hours per day for 7 consecutive days.)
* After percutaneous endoscopic gastrostomy
* Alanine Transaminase (ALT) or Aspartate Transaminase (AST): at least 3 times the upper limit of normal
* Abnormal creatinine or urea nitrogen
* Severe cardiac disease, pulmonary disease, hematic disease, autoimmune disease, mental disease, dementia and substance abuse
* History of malignancy
* History of intracranial hemorrhage
* History of severe bleeding of digestive tract, lungs, nose and skin
* Allergic to fasudil
* Participating in other clinical studies or using other investigational drugs at present

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-03 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
The slope of decline of the ALS Functional Rating Scale-Revised (ALSFRS-R) score | Month 3, 6

SECONDARY OUTCOMES:
Survival time | 2 years

OTHER OUTCOMES:
Forced Vital Capacity | Baseline, Month 3 and 6
SF-36 | Baseline, Month 3 and 6
Cognitive function | Baseline, Month 3 and 6
  verbal fluency and Frontal Behavioral Inventory Scale (FBI)
Safety Labs | Baseline, Month 0.5, 3, 3.5, 6
  blood test including blood RT, liver function, renal function, serum electrolyte, myocardial enzyme, glucose and coagulation function
Adverse Events | Month 0.5, 3, 3.5, 6

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, MD, PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China